CLINICAL TRIAL: NCT00435526
Title: Protective Efficacy of Orally Delivered Bovine Milk Immunoglobulin (BIgG) Specific for the Minor CFA/I Fimbrial Adhesin CfaE Against Challenge With H10407 Enterotoxigenic E. Coli (ETEC) Strain Expressing CFA/I
Brief Title: Efficacy of Anti-CFA/I and CfaE Bovine Milk Immunoglobulin Against Challenge With H10407 ETEC Expressing CFA/I
Acronym: BIgGI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Naval Medical Research Center (U.S. Federal Agency); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: CIR 218; HMJF Sub Award # 0000090523
Record Dates: First submitted 2007-02-13; First posted 2007-02-15 (Estimated); Last update posted 2007-02-15 (Estimated); Status verified 2007-02

CONDITIONS: Diarrhea
Keywords: traveler's diarrhea; ETEC diarrhea; passive immunization; bovine milk prophylaxis
MeSH Terms: conditions — Diarrhea

INTERVENTIONS:
Biological: anti-CFA/I bovine IgG, and anti-CfaE bovine IgG

SUMMARY:
The purpose of this study is to assess anti-CFA/I and anti-CfaE BIgG safety and to determine protective efficacy of anti-CFA/I and anti-CfaE BIgG against diarrhea after challenge with H10407, a CFA/I-expressing ETEC strain.

DETAILED DESCRIPTION:
This is a Randomized, double-blinded, placebo-controlled trial involving up to 33 subjects. Subjects will be randomized into one of the following three groups.

Group N Product

1. 10 BIgG anti-CFA/I
2. 10 BIgG anti-CfaE
3. 10 LactoFree® Lipil®

Volunteers will receive the test article three times daily following meals beginning 2 days prior to oral ETEC challenge (strain H10407). Test article will be administered for a total of 7 days. Monitoring procedures will assess volunteer safety, the primary endpoint (diarrhea), stool microbiology (H10407 excretion), and ETEC-specific immunology. All volunteers will receive antibiotic treatment (ciprofloxacin, trimethoprim-sulfamethoxazole or amoxicillin) starting 5 days after ETEC challenge or sooner based on pre-defined clinical criteria. Follow-up visits for 2 weeks post-discharge will monitor safety and immunological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 45 years of age.
* General good health, without significant medical illness, abnormal physical examination findings or clinical laboratory abnormalities as determined by principal investigator.
* Demonstrate comprehension of the protocol procedures and knowledge of ETEC illness by passing a written examination (pass grade ≥ 70%)
* Willing to participate after informed consent obtained.
* Available for all planned follow-up visits.
* Negative serum pregnancy test at screening and a negative urine pregnancy test on the day of admittance to the inpatient phase for female volunteers of childbearing potential. Females of childbearing potential must agree to use an efficacious hormonal or barrier method of birth control during the study. Abstinence is acceptable. Female volunteers unable to bear children must have this documented (e.g., tubal ligation or hysterectomy).

Exclusion Criteria:

* Presence of a significant medical condition, (e.g. psychiatric conditions or gastrointestinal disease, such as peptic ulcer, symptoms or evidence of active gastritis or gastroesophageal reflux disease, inflammatory bowel disease, alcohol or illicit drug abuse/dependency), or other laboratory abnormalities which in the opinion of the investigator precludes participation in the study.
* Immunosuppressive illness or IgA deficiency (below the normal limits)
* Positive serology results for HIV, HBsAg, or HCV antibodies.
* Significant abnormalities in screening lab hematology, serum chemistry, urinalysis or EKG (EKG in volunteers ≥ 40 years), as determined by PI.
* Allergy to fluoroquinolones, trimethoprim-sulfamethoxazole, or ampicillin/penicillin (excluded if allergic to two of three).
* Abnormal stool pattern (fewer than 3 stools per week or more than 3 stools per day) on a regular basis.
* History of diarrhea in the 2 weeks prior to planned inpatient phase
* Regular use of laxatives, antacids, or other agents to lower stomach acidity (regular defined as at least weekly).
* Use of antibiotics during the 7 days before dosing or proton pump inhibitors, H2 blockers, or antacids within 48 hours of dosing.
* Travel to countries where ETEC or cholera infection is endemic (most of the developing world) within two years prior to dosing.
* History of vaccination for or ingestion of ETEC, cholera, or LT toxin.
* Stool culture (collected no more than 1 week prior to admission) positive for CFA/I + ETEC or other bacterial enteric pathogens (Salmonella, Shigella and Campylobacter).
* Use of any investigational drug or any investigational vaccine within 30 days preceding the first dose of test article, or planned use during the active study period.
* Clinical history of lactose intolerance or allergy to milk or milk products.
* Use of any medication known to affect the immune function (e.g., corticosteroids and others) within 30 days preceding the first dose of study vaccine, or planned use during the active study period.
* Inability to tolerate an over-the-counter, lactose-free, infant, powder formula suspended in 150 mL sodium bicarbonate buffer (based on requirement for frequent dosing).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30
Dates: Start 2006-03; Study Completion 2006-10

PRIMARY OUTCOMES:
Clinical diagnosis of diarrhea defined as 1 loose/liquid stool (≥ Grade 3) of >300 g OR ≥ 2 loose/liquid stools totaling ≥ 200 g during any 48-hour period within 120 hours of challenge with ETEC strain H10407.

SECONDARY OUTCOMES:
Prevention of moderate to severe diarrhea.

CONTACTS AND LOCATIONS:
Overall Officials: Robin McKenzie, M.D., Principal Investigator — Johns Hopkins School of Public
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Medicial Center, Inpatient Unit, Baltimore, Maryland
  - General Clinical Research Center, Baltimore, Maryland